CLINICAL TRIAL: NCT07090980
Title: Effects of Podcast Education on Medication Perception, Stigma Level, and Epilepsy Self-management in Epilepsy Patients.
Acronym: epilepsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Sabahattin Zaim University (Other)
Responsible Party: Principal Investigator, Gökçe Çiçek Yavaş, Principal Investigator, Istanbul Sabahattin Zaim University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 07/2023
Record Dates: First submitted 2025-06-15; First posted 2025-07-29 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Epilepsy; Stigma; Self Management; Drug Therapy
Keywords: Epilepsy, podcast, nursing, stigma, self-management, drug perception
MeSH Terms: conditions — Epilepsy; Social Stigma

STUDY DESIGN:
Intervention Model Description: Two groups were randomly assigned as the experimental and control groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): This group was played a podcast containing information about epilepsy
  Interventions: Other: epilepsy education via podcast
- control group (No Intervention): This group received routine outpatient information about epilepsy from their doctor. No additional intervention is required.

INTERVENTIONS:
Other: epilepsy education via podcast — Epilepsy education via podcast has never been provided in any clinical study in Turkey before. By providing education via podcast, we have made health education more accessible and repeatable.
  Arms: experimental group

SUMMARY:
Seventy epilepsy patients who presented to Gaziosmanpaşa Training and Research Hospital as outpatients (diagnosed at least 3 months prior, taking at least one medication, and having access to the internet) were randomly assigned to two groups. 35 patients were assigned to the experimental group, and 35 patients to the control group. All patients were asked to complete a sociodemographic form, self-management form, medication adherence form, and stigma form as pre-tests. The experimental group was exposed to an epilepsy education podcast recorded by the researcher via Spotify. The control group received routine outpatient education provided by the doctor. The same tests were repeated at 1 and 3 months, and the effectiveness of the education was evaluated. Differences between the two groups and changes over time were monitored.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer to participate in the study
* 18 years of age
* Diagnosed with epilepsy at least 3 months ago
* Taking at least one antiepileptic drug

Exclusion Criteria:

* Being diagnosed with mental retardation
* Having language and communication barriers
* Not having sufficient equipment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2024-11-25 (Actual); Primary Completion 2025-05-15 (Actual); Study Completion 2025-05-17 (Actual)

PRIMARY OUTCOMES:
first month results | 1 month result
  Members of the intervention and control groups were assessed at the initial meeting using four forms listed by the researchers: the "Patient Information Form," the "Medication Beliefs Questionnaire," the "Feeled Stigma Scale," and the "Self-Management Scale." The control group received routine outpatient clinic education, while the patient group, designated as the intervention group, received education via a six-part podcast containing information about the epilepsy system for approximately 25 people. At the end of the training, both groups were assessed using the same four forms at the end of the first and third months.

SECONDARY OUTCOMES:
third month result | three months
  Members of the intervention and control groups were assessed at the initial meeting using four forms listed by the researchers: the "Patient Information Form," the "Medication Beliefs Questionnaire," the "Feeled Stigma Scale," and the "Self-Management Scale." The control group received routine outpatient clinic education, while the patient group, designated as the intervention group, received education via a six-part podcast containing information about the epilepsy system for approximately 25 people. At the end of the training, both groups were assessed using the same four forms at the end of the first and third months.

CONTACTS AND LOCATIONS:
Locations (1):
- Gaziosmanpaşa Eğitim ve Araştırma Hastanesi, Istanbul, gaziosmanpaşa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Personal data will not be shared for the purpose of protecting personal data.